CLINICAL TRIAL: NCT05272631
Title: Depuy Synthes Lower Extremity Shaft Nail Registry (RFN-Advanced™ Retrograde Femoral Nailing System/ TN-Advanced™ Tibial Nailing System)
Brief Title: Depuy Synthes Lower Extremity Shaft Nail Registry
Status: Completed | Type: Observational
Sponsor: DePuy Synthes Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DST202103; DST202103 (Other: DePuy Synthes Products, Inc.)
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Femoral Fractures; Tibial Fractures
MeSH Terms: conditions — Femoral Fractures; Tibial Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Retrograde Femoral Nail Advanced (RFNA) Cohort: Participants with a distal femur or femoral shaft fracture or who require revision due to a malunion or nonunion will undergo surgery with RFNA based on surgeon's decision and the site's standard of care (SOC). Participants with impending pathologic fracture are also included.
  Interventions: Device: Retrograde Femoral Nail Advanced
- Tibial Nail Advanced (TNA) Cohort: Participants with open or closed, proximal, distal or shaft fractures of the tibia, or who require revision due to a malunion or nonunion will undergo surgery with TNA based on surgeon's decision and the site's SOC.
  Interventions: Device: Tibial Nail Advanced

INTERVENTIONS:
Device: Retrograde Femoral Nail Advanced — No drug will be given as part of this study. Participant will undergo surgery with RFNA based on the surgeon's decision and the site's SOC.
  Groups: Retrograde Femoral Nail Advanced (RFNA) Cohort
Device: Tibial Nail Advanced — No drug will be given as part of this study. Participant will undergo surgery with TNA based on the surgeon's decision and the site's SOC.
  Groups: Tibial Nail Advanced (TNA) Cohort

SUMMARY:
The purpose of this post-market registry is to monitor the clinical safety and performance (union rates and time to union) of two DePuy Synthes lower extremity shaft nails: RFN-Advanced Retrograde Femoral Nailing System (RFNA) and TN-Advanced Tibial Nailing System (TNA) in participants who have experienced femoral or tibial fractures, respectively, requiring fixation and stabilization or who require a revision due to a malunion or a nonunion.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature adults age greater than or equal to (>=) 22 years (Retrograde Femoral Nail Advanced [RFNA], Tibial Nail Advanced [TNA]) and adolescents 12-21 years of age in which the growth plates have fused (TNA only)
* Participant receives an RFNA and/or TNA based on a diagnosis of open or closed, unilateral or bilateral femoral shaft or distal femur fracture (RFNA); unilateral or bilateral tibial fracture (TNA); revision of malunion or nonunion of previous fracture, or impending pathologic fracture (RFNA only) that will be treated operatively as part of standard of care. In addition, the following will be included: a) RFNA only: femoral shaft or distal femur fracture can be periprosthetic (PPFx) fracture after total or unicondylar knee arthroplasty, or total or hemi hip arthroplasty requiring nail osteosynthesis
* Participant (legally authorized representative if participant is a minor) voluntarily signs the Institutional Review Board (IRB)/ Ethics committee (EC) approved consent form
* Participant must be able to read and understand questions and responses in an available translated language for patient reported outcomes (PROs)

Exclusion Criteria:

* Participation in any other medical device or medicinal product study within the previous month. Participation in observational studies is allowed
* In the opinion of the Principal Investigator, participant is unable to comply with the requirements of the Registry
* Participant has known allergies to implant components

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes adults 22 years of age or older, (Retrograde Femoral Nail Advanced [RFNA], Tibial Nail Advanced [TNA]) or adolescents 12-21 years of age in which the growth plates have fused (TNA only) who will undergo surgery for fixation and stabilization of a tibia, femoral shaft or distal femur fracture, or who require a revision due to a malunion or a nonunion, with either the TNA (tibia) or RFNA (femoral shaft or distal femur).
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Time to Union | Up to Week 56
  Time to union will be reported. Union is defined as a combination of radiographic and clinical assessment, where union will be considered achieved based on radiographic images, and no pain at the fracture site indicative of nonunion.
Number of Participants with Union (Healing) | Up to Week 56
  Number of participants with union (healing) will be reported. Union is defined as a combination of radiographic and clinical assessment, where union will be considered achieved based on radiographic images, and no pain at the fracture site indicative of nonunion.

SECONDARY OUTCOMES:
Pain Visual Analogue Scale (VAS) Score | From Week 6 up to Week 52
  The VAS is a 100 point one-dimensional line anchored on either end by verbal descriptors ranging from " 0=no pain" to "100=worst pain you can imagine". The higher score indicates greater pain intensity.
Short Form 12-Item Health Survey (SF-12) Questionnaire Score | From Week 6 up to Week 52
  The SF-12 volume-2 is a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). Mental health-related scales include Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH). For each of the 8 domains, the questions are coded, added and transformed on a scale that ranges from 0 (the worst health status for that dimension) to 100 (the best health status).
Quality of Life as Assessed by European Quality of Life (EuroQoL) 5-Dimensions 5-Levels (EQ-5D-5L) Questionnaire Score: EQ-5D Descriptive System | From Week 6 up to Week 52
  EQ-5D-5L is a standardized instrument that was designed for self-completion. EQ-5D-5L consist of EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This decision results in a 1-digit number that expresses the level selected for that dimension. The scores are applied to population-specific valuations of health states to result in a single index value. The health index scores generally range from less than 0 to 1 with higher scores indicating higher health utility.
Quality of Life as Assessed by EQ-5D-5L Questionnaire Score: EQ VAS | From Week 6 up to Week 52
  EQ-5D-5L is a standardized instrument that was designed for self-completion. EQ-5D-5L consist of EQ-5D descriptive system and the EQ VAS. The EQ VAS records the participant's self-rated health on a vertical visual analogue scale from 0 to 100, where 0 indicate 'The best health you can imagine' and 100 indicate 'The worst health you can imagine'.
Weight Bearing Status | From Week 2 up to Week 52
  Weight bearing status will be categorized as weight-bearing as tolerated (WBAT), limited weight-bearing up to half of the body weight, and no weight bearing.
Mobility Assessment | Up to Week 56
  Mobility assessment including ambulatory/unaided, ambulatory with cane, ambulatory with walker and nonambulatory will be reported.
Number of Participants with Revision Surgery | From Week 2 up to Week 52
  Number of participants with revision surgery will be reported. It includes the surgery following the index surgery that involves adjustment, modification, removal or replacement of the implanted device or other associated devices used to treat the fracture (nail, screws, endcaps, locking attachment washer [LAW] [Retrograde Femoral Nail Advanced {RFNA} only] or condylar nut and nut and screw washers [RFNA only]).
Number of Participants with Reoperation | From Week 2 up to Week 52
  Number of participants with reoperation will be reported. It is defined as a second operation at the fracture site(s) after the index surgery that does not include adjustment, modification, removal or replacement of the implanted device.

CONTACTS AND LOCATIONS:
Overall Officials: DePuy Synthes Products, Inc. Clinical Trial, Study Director — DePuy Synthes Products, Inc.
Locations (8):
- United States (8):
  - Orthopedic Research Foundation, Inc, Indianapolis, Indiana
  - Michigan Medicine; University of Michigan, Ann Arbor, Michigan
  - University of Missouri, Columbia, Missouri
  - Duke University, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - JPS Health Network, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Beak P, Moudhgalya S, Anderson T, Hing CB. Painful locking screws with tibial nailing, an underestimated complication. Eur J Orthop Surg Traumatol. 2019 Dec;29(8):1795-1799. doi: 10.1007/s00590-019-02501-8. Epub 2019 Jul 16. PMID 31312954
- [Background] Byun SE, Shon HC, Park JH, Oh HK, Cho YH, Kim JW, Sim JA. Incidence and risk factors of knee injuries associated with ipsilateral femoral shaft fractures: A multicentre retrospective analysis of 429 femoral shaft injuries. Injury. 2018 Aug;49(8):1602-1606. doi: 10.1016/j.injury.2018.06.006. Epub 2018 Jun 4. PMID 29887503
- [Background] Capone A, Congia S, Civinini R, Marongiu G. Periprosthetic fractures: epidemiology and current treatment. Clin Cases Miner Bone Metab. 2017 May-Aug;14(2):189-196. doi: 10.11138/ccmbm/2017.14.1.189. Epub 2017 Oct 25. PMID 29263732
- [Background] Cereijo C, Attum B, Rodriguez-Buitrago A, Jahangir AA, Obremskey W. Intramedullary Nail Fixation of Tibial Shaft Fractures: Suprapatellar Approach. JBJS Essent Surg Tech. 2018 Sep 12;8(3):e24. doi: 10.2106/JBJS.ST.17.00063. eCollection 2018 Sep 28. PMID 30588369
- [Background] Court-Brown CM, Caesar B. Epidemiology of adult fractures: A review. Injury. 2006 Aug;37(8):691-7. doi: 10.1016/j.injury.2006.04.130. Epub 2006 Jun 30. PMID 16814787
- [Background] Court-Brown CM. The epidemiology of fractures and dislocations. In: Court-Brown CM, Heckman JD, Mcqueen MM, et al, eds. Rockwood and Green's Fractures in Adults. 8th ed. Philadelphia, PA: Wolters Kluwer Health; 2015:59-108
- [Background] EQ-5D-5L User Guide, EuroQol Research Foundation 2019; Version 3.0 Updated Sept. 2019
- [Background] Finkemeier, C et al. (2020a, August 30). RFN-Advanced Retrograde Femoral Nailing System. https://approvedsolutions.aofoundation.org/approvedsolutionsfolder/2020/rfn-advancedretrograde- femoral-nailing-system#tab=details TN- Advanced Tibial Nailing System https://approvedsolutions.aofoundation.org/approvedsolutionsfolder/2020/t -advanced-tibialnailing- system#tab=details;
- [Background] Finkemeier, C et al. (2020b, November 24) Advanced Nailing System. AO Innovations Magazine 2020. https://issuu.com/aofoundation/docs/aoe_tc_innovations_24_11_2020_final
- [Background] He GC, Wang HS, Wang QF, Chen ZH, Cai XH. Effect of minimally invasive percutaneous plates versus interlocking intramedullary nailing in tibial shaft treatment for fractures in adults: a meta-analysis. Clinics (Sao Paulo). 2014;69(4):234-40. doi: 10.6061/clinics/2014(04)03. PMID 24714830
- [Background] Lee C, Zoller SD, Perdue PW Jr, Nascone JW. Pearls and Pitfalls With Intramedullary Nailing of Proximal Tibia Fractures. J Am Acad Orthop Surg. 2020 Jan 15;28(2):66-73. doi: 10.5435/JAAOS-D-18-00765. PMID 31884503
- [Background] Meena RC, Meena UK, Gupta GL, Gahlot N, Gaba S. Intramedullary nailing versus proximal plating in the management of closed extra-articular proximal tibial fracture: a randomized controlled trial. J Orthop Traumatol. 2015 Sep;16(3):203-8. doi: 10.1007/s10195-014-0332-9. Epub 2015 Jan 15. PMID 25588847
- [Background] Oak SR, Strnad GJ, Bena J, Farrow LD, Parker RD, Jones MH, Spindler KP. Responsiveness Comparison of the EQ-5D, PROMIS Global Health, and VR-12 Questionnaires in Knee Arthroscopy. Orthop J Sports Med. 2016 Dec 17;4(12):2325967116674714. doi: 10.1177/2325967116674714. eCollection 2016 Dec. PMID 28210645
- [Background] Rodriguez EK, Boulton C, Weaver MJ, Herder LM, Morgan JH, Chacko AT, Appleton PT, Zurakowski D, Vrahas MS. Predictive factors of distal femoral fracture nonunion after lateral locked plating: a retrospective multicenter case-control study of 283 fractures. Injury. 2014 Mar;45(3):554-9. doi: 10.1016/j.injury.2013.10.042. Epub 2013 Nov 4. PMID 24275357
- [Background] Yoon BH, Park IK, Kim Y, Oh HK, Choo SK, Sung YB. Incidence of nonunion after surgery of distal femoral fractures using contemporary fixation device: a meta-analysis. Arch Orthop Trauma Surg. 2021 Feb;141(2):225-233. doi: 10.1007/s00402-020-03463-x. Epub 2020 May 9. PMID 32388648